CLINICAL TRIAL: NCT02619448
Title: Pilot Study of the Safety and Feasibility of Administering Concurrent Chemotherapy and Accelerated Hypofractionated Radiation Therapy in the Treatment of Medically Inoperable T2A-T4 N0 Non-small Cell Lung Cancer.
Brief Title: Concurrent Chemotherapy Plus HFR Radiation Therapy in Inoperable NSCLC
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 665895
Record Dates: First submitted 2015-03-16; First posted 2015-12-02 (Estimated); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: inoperable; Solitary [T1bN0, T2aN0, T2bN0] lesion measuring 2-7 cm
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy with hypofractionated RT (Experimental): Carboplatin AUC 2 + Paclitaxel 50 mg/m2 given weekly x 4 concurrently with radiation therapy (70 Gy in 20 fractions) over 4 weeks
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Radiation: 70 Gy in 20 fractions over 4 weeks

INTERVENTIONS:
Drug: Carboplatin — chemotherapy
  Other Names: Paraplatin
Drug: Paclitaxel — chemotherapy
  Other Names: taxol
Radiation: 70 Gy in 20 fractions over 4 weeks — accelerated hypofractionated RT

SUMMARY:
The standard treatment for patients with Non-Small Cell Lung Cancer (NSCLC) and clinically negative lymph nodes remains surgery per current guidelines. Five year survival for patients with stage I non-small cell lung cancer is generally greater than 50% after surgery. Many of these patients have heart and lung issues or other diseases which keep them from undergoing curative surgery. Studies have shown that majority of these patients die from their cancer and not from their other diseases. This is the reason for treating early stage lung cancer patients with definitive therapy, when they cannot have surgery. This study will enroll twelve subjects to evaluate the side effects of this treatment, and decide if it is a good option for the patients that cannot have surgery.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer related deaths for both men and women in the United States. In 2014 the estimated number of new lung cancer cases in the United States is 224,210. Approximately 159,260 people are estimated to die from lung cancer in 2014. Non-small cell lung cancer (NSCLC) constitutes 80% of all lung cancer cases. The standard treatment for patients with NSCLC and clinically negative lymph nodes remains surgery per NCCN guidelines. Five year survival for patients with stage I non-small cell lung cancer is generally greater than 50% after surgical resection with lobectomy. A significant number of these patients have cardio-pulmonary or other co-morbidities which preclude them from undergoing curative surgery. Studies have shown that majority of these patients die from their cancer and not from their co-morbidities. This forms the rationale for treating medically inoperable early stage lung cancer patients with definitive therapy.

Treatment with radiotherapy (RT) has been the standard option for patients unable to undergo surgery. Radiation alone leads to slightly better outcomes but still not equivalent to surgery with 60-70% local failure with conventional fractionated radiotherapy over several weeks. The development of three-dimensional conformal radiotherapy (3DCRT) has allowed for more focused treatment while avoiding nearby normal tissue resulting in improved disease specific survival but overall survival is still poor.

There is currently no data supporting the use of chemotherapy in the medically inoperable group either in an adjuvant setting or concurrently with RT in those with early stage lung cancer. In patients with unresectable Stage IIIA and IIIB NSCLC, combined chemo-RT has been proven to be superior to RT alone. Two randomized studies that compared concurrent versus sequential chemo-radiotherapy found that the concurrent approach provides superior outcomes. However this approach has not been studied in early stage lung cancer in the medically inoperable group. The medically inoperable patient cohort often does not undergo surgical staging, which increases the odds that they harbor occult regional disease. Chemotherapy given concurrently with radiation will act as a radiosensitizer and improve local disease control and could decrease rate of distant metastases. It is possible that the medically inoperable population also experience more side effects due to their co-morbidities and poor performance status. Hence there is a need to determine if concurrent chemoradiation is feasible and tolerable in the medically inoperable patients. The main side effect associated with concurrent chemoradiation in stage III NSCLC is esophagitis. This arises due to effect of radiation therapy to the regional lymph node (LN). The investigators' study population with early stage lung cancer has no nodal involvement. Hence, the investigators do not anticipate esophagitis being a major side effect in the researchers' study.

There is recent data for adjuvant chemotherapy in the medically operable group. Data from the Lung Adjuvant Cisplatin Evaluation (LACE) showed with a median follow-up time of 5.2 years, the overall HR of death was 0.89 (95% CI, 0.82 to 0.96; P = .005), corresponding to a 5-year absolute benefit of 5.4% from chemotherapy. A similar trial evaluating the role of sequential chemotherapy after stereotactic body radiation therapy (SBRT) in the medically inoperable population was attempted at the investigators' institution but was closed due to poor accrual. Hence, the investigators are looking at the role of concurrent chemo-RT in this population.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically or cytologically proven diagnosis of non-small cell lung carcinoma.
* Solitary [T1bN0M0, T2aN0M0, T2bN0M0] lesion measuring 2-7cm in size. Staging is per AJCC 7th edition of TNM classification.
* Patient must meet criteria for receipt of hypofractionated radiation therapy
* Medically inoperable pulmonary status, cardiac status, or other serious co-morbidity, or patient refusal of primary surgery for lung cancer.
* ECOG Performance status of 0-2.
* Patients may have prior treatment for lung cancer based on the following criteria:

  1. Surgical resection is allowed if surgery was > 12 months ago.
  2. Patients treated with prior radiation are eligible if radiation was > 12 months ago and there is no evidence of progression and if the lesion is in a different lobe.
  3. Prior chemotherapy if > 18 months ago

Exclusion Criteria:

* Node positive or metastatic disease.
* Other active malignancy (specifically, risk of recurrence in 3 years estimated to be greater than 50%) except for non-melanoma skin cancer, in-situ cervical carcinoma (CIN), or low-risk prostate carcinoma on active surveillance are to be excluded.
* Inability to receive systemic therapy or radiation therapy per protocol.
* Inability to fulfill requirements of the protocol.
* Any co-morbidity or condition which, in the opinion of the investigator, may interfere with the assessments and procedures of this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-12; Primary Completion 2024-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Toxicity as measured using the National Cancer Institute's Common Terminology Criteria for Adverse Events | 24 months
  Specifically grade 3+ toxicity associated with the treatment will be summarized by grade and type.

SECONDARY OUTCOMES:
Radiographic response as measured by PET/CT | 24 months
Local progression as measured by PET/CT | 24 months
Regional progression as measured by PET/CT | 24 months
Distant progression as measured by PET/CT | 24 months
Time to overall progressions as measured by PET/CT | 24 months
Overall survival as determined by patient contact | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mix, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States